CLINICAL TRIAL: NCT04655326
Title: Assessment of Customized Probiotic Therapy for Children and Adults With Autism Spectrum Disorder
Brief Title: Probiotic Therapy for Children and Adults With Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Sun Genomics (Unknown)
Responsible Party: Principal Investigator, James B Adams, President's Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00012299
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — crataegus extract

STUDY DESIGN:
Intervention Model Description: Each participant receives a customized probiotic based on the results of the measurement of their gut microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Each participant receives a customized probiotic based on the results of the test of their microbiota
  Interventions: Biological: Flore

INTERVENTIONS:
Biological: Flore — personalized blend of GRAS approved probiotic strains, prebiotics, and botanicals

SUMMARY:
This is a study of the effect of a customized probiotic on children and adults with autism, including effects on autism symptoms and gastrointestinal symptoms.

DETAILED DESCRIPTION:
SunGenomics provides its customers with a customized probiotic based on an analysis of the microbiota in their stool samples. Customers who have autism spectrum disorders are invited to participate in this study by completing several questionnaires about their medical history, diet, autism symptoms, and gastrointestinal symptoms before taking the probiotic, and to repeat those questionnaires approximately 3 months later. This is effectively an open-label study.

ELIGIBILITY:
Inclusion Criteria:

1. New client of Sun Genomics (has applied for testing and treatment, but not yet begun treatment)
2. Diagnosis of ASD (initially based on self-report of ASD diagnosis by appropriate medical professional, and then verified by an evaluation of the Social Responsiveness Scale (SRS-2) by ASU staff.
3. Children and adults ages 2.5-75 years

Exclusion Criteria:

1. Antibiotic use in the last two months (not counting topical antibiotics)
2. Any changes in medications, nutritional supplements, therapies, in the last two months, or any plans to change them during the first 3 months of probiotic treatment.

Ages: 30 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Parent Global Impressions of Autism | change in score between baseline and 3 months
  questionnaire which assesses 20 different autism-related symptoms on a 7-point scale

SECONDARY OUTCOMES:
Social Responsiveness Scale | change in score between baseline and 3 months
  A questionnaire about social skills, where higher scores suggest more severe autism. Scores range from 0 to 195, with higher scores indicating more severe problems.
Gastrointestinal Symptom Rating Scale | change in score between baseline and 3 months
  A questionnaire which evaluates 15 gastrointestinal symptoms on a severity scale from 1 (none) to 7 (severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: link to official study ad — https://autism.asu.edu/research-studies